CLINICAL TRIAL: NCT05918419
Title: Neoadjuvant Chemoradiation Plus Serplulimab in Patients With Locally Advanced Adenocarcinoma of Gastroesophageal Junction: a Single-arm,Open-label，Phase II Clinical Study
Brief Title: Efficacy and Safety of Neoadjuvant Chemoradiation Plus Serplulimab in Patients With Locally Advanced Adenocarcinoma of Gastroesophageal Junction
Acronym: SNACRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-GEJ-IIT
Record Dates: First submitted 2023-06-04; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-01

CONDITIONS: Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemoradiation (Experimental): neoadjuvant chemoradiation plus PD-1 antibody (Serplulimab) Intervention: Drug: Neoadjuvant chemoradiation plus PD-1 antibody(Serpluimab)
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — PD-1 antibody

SUMMARY:
Investigators conduct the clinical trial to further explore the efficacy and safety of Neoadjuvant chemoradiation Plus Serpluimab in Patients with locally advanced Adenocarcinoma of Gastroesophageal Junction

DETAILED DESCRIPTION:
1. Target population: patients with locally advanced adenocarcinoma of Gastroesophageal Junction (cT3-4aN+M0).
2. Primary objective: pathological complete remission (pCR) rate of neoadjuvant chemoradiation plus Serpluimab in patients with locally advanced Adenocarcinoma of Gastroesophageal Junction
3. Patients will be given the perioperative treatment as below once recruited:

   induction chemotherapy ：Serplulimab 300mg iv.gtt d1+Oxaliplatin130mg/m2 iv.gtt d1,+S1 40mg/m2 p.o.b.i.d. d1~d14（up to 60mg) .Every three weeks for one cycle.

   After the induction chemotherapy，concurrent chemoradiation will be strated：Serplulimab 300mg iv.gtt d1,+Oxaliplatin100mg/m2 iv.gtt d1+S1 40mg/m2 p.o.b.i.d.

   d1~d14(up to 60mg), every three weeks , the total of two cycles . Radiation total dose: 45Gy/25F, 1.8Gy/d. Resectable patients will receive D2 resection After 6-8weeks Neoajuvant therapy
4. Number of subjects: 35 patients. Number of centers: 1 site(Peking Union Medical College Hospital)

ELIGIBILITY:
Inclusion Criteria:

1. histologically documented adenocarcinoma of Gastroesophageal Junction.
2. clinically diagnosed stage T3-4aN+M0 according to ultrasound endoscopy or enhanced CT/MRI scan.
3. Male or female. Age ≥ 18 years and ≤75 years.
4. surgeons participating in this study consider the lesion a resectable one.
5. ECOG 0~1
6. Physical condition and adequate organ function to ensure the success of abdominal surgery.
7. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥90g/L.
8. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN . ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.
9. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 60 ml/min.
10. Adequate coagulation function: INR/PT≤ 1.5 x ULN, aPTT≤ 1.5 x ULN.
11. No serious concomitant disease that will threaten the survival of patients to less than 5 years.
12. Written (signed) informed consent.
13. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
14. Female patients should not be pregnant or breast feeding.
15. PD-L1 assessment

Exclusion Criteria:

1. patients with distant metastasis or unresectable primary lesion.
2. patients with T1, T2 lesion according to CT/MRI or ultrasound endoscopy.
3. history of chemo, radiation, immune therapy or radical resection for the GEJ.
4. patients with active autoimmune disease or history of refractory autoimmune disease.
5. patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured locally tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ.
6. uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment.
7. patients who have digestive tract bleeding in 2 weeks before recruitment or with high risk of bleeding.
8. perforation / fistula of GI tract in 6 months before recruitment.
9. patients with upper GI tract obstruction or functional abnormality or malabsorption syndrome, which can affect absorption of S-1.
10. losing over 20% body weight in 2 months before recruitment.
11. pulmonary disease history: interstitial pulmonary disease, non-infective pneumonitis, pulmonary fibrosis, acute pulmonary disease.
12. uncontrollable systemic diseases, including diabetes, hypertension, etc.
13. severe chronic or active infections in need of systemic antibacterial, antifungal, or antiviral treatment, including TB or HIV, etc.
14. patients with untreated chronic hepatitis B or HBV DNA over 500 IU/ml or positive HCV RNA.
15. patients with any cardiovascular risk factors below:

    1. cardiac chest pain occurring in 28 days before recruitment, defined as moderate pain that limits daily activity.
    2. pulmonary embolism with symptoms occurring in 28 days before recruitment.
    3. acute myocardial infarction occurring in 6 months before recruitment.
    4. any history of heart failure reaching grade 3/4 of NYHA in 6 months before recruitment.
    5. ventricular arrhythmias of Grade 2 or grater in 6 months before recruitment, or accompanied by supraventricular tachyarrhythmias requiring medical treatment.
    6. cerebrovascular accident within 6 months before recruitment.
16. patients with peripheral neuropathy NCI CTC AE grade 1, except those with only deep tendon reflex disappearing.
17. moderate or severe renal injury [creatinine clearance rate≤50 ml/min (according to Cockroft & Gault equation)], or Scr>1.5 x ULN.
18. dipyrimidine dehydrogenase (DPD) deficiency.
19. allergic to any drug in this study.
20. history of allogeneic stem cell transplantation or organ transplantation.
21. use of steroids (dosage>10mg/d prednisone) or other systemic immune suppressive therapy in 14 days before recruitment, except patients treated with regimens below: a. steroids for hormone replacement (dosage>10mg/d prednisone); b. steroids for local application with little systemic absorption; c. short -term (≤ 7 days) steroids for preventing allergy or vomiting.
22. vaccinated with live vaccine in 4 weeks before recruitment.
23. receiving immune (interleukin, interferon, thymin) treatment or treatment of other trials in 28 days before recruitment.
24. receiving palliative radiation in 14 days before recruitment.
25. history of anti PD-1, PD-L1, PD-L2 or any other specific T cell co-stimulation or checkpoint pathway targeted treatment.
26. receiving operation in 28 days before recruitment, only if the operation is a minimally invasive one e.g. PICC.
27. for patients with uncontrolled epilepsy, CNS diseases or history of mental disorder, researchers should evaluate whether their diseases will impede their signing of informed consent or compliance of treatment.
28. existing of potential situation which will impede drug administration or affect toxicity analysis or alcohol/ drug abuse.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete regression (pCR) rate | 3 months after the last subject participating in
  pathological complete remission (pCR) rate of Neoadjuvant Chemoradiation Plus Serplulimab in Patients With Locally Advanced Adenocarcinoma of Gastroesophageal Junction

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China